CLINICAL TRIAL: NCT03066102
Title: Muscle Fatigue and Scapular Sensorimotor System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yi-Fen Shih, Associate Professor, National Yang Ming Chiao Tung University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: YM105067E
Record Dates: First submitted 2017-02-16; First posted 2017-02-28 (Actual); Results first posted 2019-07-15 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Muscle; Fatigue
Keywords: sensorimotor system; scapular joint position sense; fatigue
MeSH Terms: conditions — Fatigue | interventions — Muscle Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: muscle fatigue — Modified push-up plus exercise:
  the participants first supported by both knees and the single elbow, and then performed sustained scapular protraction for three minutes with ten repetitions in males and two minutes with five repetitions in females with forty-five seconds rest between.

SUMMARY:
The aims of this study are to investigate the effects of scapular muscle fatigue on scapular joint position sense and neuromuscular performance (scapular muscle strength, the kinematics data and muscle activity of shoulder during scaption (arm elevation in the scapular plane)). The investigators hypothesize that scapular muscle fatigue would increase scapular reposition error and affect neuromuscular performance of the scapular during scaption.

ELIGIBILITY:
Inclusion Criteria:

* no shoulder, cervical, and thoracic spine pain within six months
* negative for subacromial impingement test
* normal range of motion of glenohumeral joint

Exclusion Criteria:

* history of dislocation, fracture, or surgery of shoulder joint
* history of central nervous system disorder, rheumatoid arthritis, shoulder osteoarthritis, or cervical radiculopathy

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-08-11 (Actual); Study Completion 2018-03-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Yang Ming University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Fatigued Group: Subjects held in a modify pushup plus position. Like an all four position, subjects hold with right arm with elbow flexion and full shoulder protraction. Male subjects had to hold three minutes for ten repetitions, and female subjects were two minutes for five repetitions. There was thirty second rest between repetitions. The end of fatigue task was: subjects finished all the repetition, or could not do one more repetition. Female subjects could do more than five repetitions if they felt ok, and the maximum repetitions were ten. The muscle activation of upper trapezius, lower trapezius, and serratus would record for analysis of median frequency. As long as finished fatigue task, the post measurements would start.
Period: Overall Study
Arm/Group | Fatigued Group
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Fatigued Group: the only group in this study, and every subjects took the fatigued task
Arm/Group | Fatigued Group
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.5 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
height [Mean (Standard Deviation); unit: centimeters] | 167.57 (8.29)
weight [Mean (Standard Deviation); unit: kilograms] | 59.30 (8.53)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Scapular Proprioception
Description: Test the ability of active re-position the scapula from neutral to 90% range of protraction, and elevation.
Time Frame: through fatigue intervention completion, an average of 20 minutes in female subjects and 40 minutes in male subjects
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Fatigued Group
Number analyzed (Participants) | 30
centimeters
  elevation task: pre-test | -0.48 (0.88)
  elevation task: post-test | -0.19 (1.05)
  protraction task: pre-test | -0.37 (0.61)
  protraction task: post-test | -0.32 (0.73)
Statistical Analysis 1: Comparison: Fatigued Group; The effects of muscle fatigue on reposition error of scapular elevation. Muscle fatigue would increase reposition error during scapular elevation. One-way repeated measures analysis of variance; Test type: Other; p = 0.227, ANOVA — The level of statistical significance was set at P < 0.05
Statistical Analysis 2: Comparison: Fatigued Group; The effects of muscle fatigue on reposition error of scapular protraction. Muscle fatigue would increase reposition error during scapular protraction. One-way repeated measures analysis of variance; Test type: Other; p = 0.764, ANOVA — The level of statistical significance was set at P < 0.05

2. Primary Outcome: Change From Baseline in Muscle Activation During Scapular Proprioception
Description: Test the ability of muscle activation (upper trapezius, lower trapezius, and serratus anterior) during active re-position the scapula from neutral to 90% range of protraction, and elevation.
  Muscle activation during active re-position would divide into muscle activation during maximum voluntary isometric contraction (MVIC), present in percent.
Time Frame: through fatigue intervention completion, an average of 20 minutes in female subjects and 40 minutes in male subjects
Measure: Mean (Standard Deviation); unit: percentage of MVIC
Arm/Group | Fatigued Group
Number analyzed (Participants) | 30
percentage of MVIC
  serrates anterior during elevation: pre-test | 18.48 (11.05)
  serrates anterior during elevation: post-test | 26.34 (18.76)
  serrates anterior during protraction: pre-test | 15.22 (12.54)
  serrates anterior during protraction: post-test | 27.41 (38.03)
  upper trapezius during elevation: pre-test | 45.17 (20.18)
  upper trapezius during elevation: post-test | 52.46 (53.62)
  upper trapezius during protraction: pre-test | 8.28 (7.11)
  upper trapezius during protraction: post-test | 10.49 (13.77)
  lower trapezius during elevation: pre-test | 3.51 (1.97)
  lower trapezius during elevation: post-test | 3.51 (2.17)
  lower trapezius during protraction: pre-test | 6.41 (5.11)
  lower trapezius during protraction: post-test | 5.59 (4.58)
Statistical Analysis 1: Comparison: Fatigued Group; The effects of muscle fatigue on muscle activation of upper trapezius during scapular elevation. Muscle fatigue would change muscle activation during proprioception task. One-way repeated measures analysis of variance; Test type: Other; p = 0.413, ANOVA — The level of statistical significance was set at P < 0.05
Statistical Analysis 2: Comparison: Fatigued Group; The effects of muscle fatigue on muscle activation of lower trapezius during scapular elevation. Muscle fatigue would change muscle activation during proprioception task. One-way repeated measures analysis of variance; Test type: Other; p = 0.984, ANOVA — The level of statistical significance was set at P < 0.05
Statistical Analysis 3: Comparison: Fatigued Group; The effects of muscle fatigue on muscle activation of serratus anterior during scapular elevation. Muscle fatigue would change muscle activation during proprioception task. One-way repeated measures analysis of variance; Test type: Other; p = 0.006, ANOVA — The level of statistical significance was set at P < 0.05
Statistical Analysis 4: Comparison: Fatigued Group; The effects of muscle fatigue on muscle activation of upper trapezius during scapular protraction. Muscle fatigue would change muscle activation during proprioception task. One-way repeated measures analysis of variance; Test type: Other; p = 0.154, ANOVA — The level of statistical significance was set at P < 0.05
Statistical Analysis 5: Comparison: Fatigued Group; The effects of muscle fatigue on muscle activation of lower trapezius during scapular protraction. Muscle fatigue would change muscle activation during proprioception task. One-way repeated measures analysis of variance; Test type: Other; p = 0.096, ANOVA — The level of statistical significance was set at P < 0.05
Statistical Analysis 6: Comparison: Fatigued Group; The effects of muscle fatigue on muscle activation of serratus anterior during scapular protraction. Muscle fatigue would change muscle activation during proprioception task. One-way repeated measures analysis of variance; Test type: Other; p = 0.037, ANOVA — The level of statistical significance was set at P < 0.05

3. Secondary Outcome: Change From Baseline in Scapular Muscle Strength
Description: use dynamometer to detect the force of maximum isometric voluntary contraction of upper trapezius, lower trapezius and serratus anterior
Time Frame: through fatigue intervention completion, an average of 20 minutes in female subjects and 40 minutes in male subjects
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Fatigued Group
Number analyzed (Participants) | 30
kilograms
  serrates anterior muscle: pre-test | 10.42 (3.92)
  serrates anterior muscle: post-test | 8.40 (3.60)
  upper trapezius muscle: pre-test | 23.39 (10.99)
  upper trapezius muscle: post-test | 20.87 (10.48)
  lower trapezius muscle: pre-test | 4.47 (2.08)
  lower trapezius muscle: post-test | 4.31 (1.89)
Statistical Analysis 1: Comparison: Fatigued Group; The effects of muscle fatigue on muscle strength of serratus anterior during maximum voluntary isometric muscle contraction. Muscle fatigue would decrease muscle strength during maximum voluntary isometric muscle contraction. One-way repeated measures analysis of variance; Test type: Other; p = 0.000085, ANOVA — The level of statistical significance was set at P < 0.05
Statistical Analysis 2: Comparison: Fatigued Group; The effects of muscle fatigue on muscle strength of upper trapezius during maximum voluntary isometric muscle contraction. Muscle fatigue would decrease muscle strength during maximum voluntary isometric muscle contraction. One-way repeated measures analysis of variance; Test type: Other; p = 0.037, ANOVA — The level of statistical significance was set at P < 0.05
Statistical Analysis 3: Comparison: Fatigued Group; The effects of muscle fatigue on muscle strength of lower trapezius during maximum voluntary isometric muscle contraction. Muscle fatigue would decrease muscle strength during maximum voluntary isometric muscle contraction. One-way repeated measures analysis of variance; Test type: Other; p = 0.382, ANOVA — The level of statistical significance was set at P < 0.05

4. Secondary Outcome: Change From Baseline in Shoulder Kinematics Data During Shoulder Elevation in the Scapular Plane
Description: use Liberty to detect the motion of spine, humerus, and scapula during shoulder elevation in the scapular plane (scaption)
Time Frame: through fatigue intervention completion, an average of 20 minutes in female subjects and 40 minutes in male subjects
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Fatigued Group
Number analyzed (Participants) | 30
degree
  posterior tilt ascending 30 degree: pre-test | 0.68 (4.79)
  posterior tilt ascending 60 degree: pre-test | 7.60 (5.75)
  posterior tilt ascending 90 degree: pre-test | 10.84 (7.43)
  posterior tilt ascending 120 degree: pre-test | 13.81 (12.22)
  posterior tilt ascending 30 degree: post-test | 0.05 (4.98)
  posterior tilt ascending 60 degree: post-test | 6.77 (5.93)
  posterior tilt ascending 90 degree: post-test | 9.53 (8.04)
  posterior tilt ascending 120 degree: post-test | 10.33 (13.40)
  posterior tilt descending 120 degree: pre-test | 11.44 (14.00)
  posterior tilt descending 90 degree: pre-test | 8.54 (7.96)
  posterior tilt descending 60 degree: pre-test | 4.02 (5.89)
  posterior tilt descending 30 degree: pre-test | -2.47 (5.09)
  posterior tilt descending 120 degree: post-test | 7.63 (14.24)
  posterior tilt descending 90 degree: post-test | 6.64 (8.61)
  posterior tilt descending 60 degree: post-test | 2.72 (6.63)
  posterior tilt descending 30 degree: post-test | -3.55 (5.41)
  internal rotation ascending 30 degree: pre-test | 11.37 (5.44)
  internal rotation ascending 60 degree: pre-test | 11.02 (5.89)
  internal rotation ascending 90 degree: pre-test | 10.68 (7.52)
  internal rotation ascending 120 degree: pre-test | 10.21 (13.57)
  internal rotation ascending 30 degree: post-test | 10.84 (5.23)
  internal rotation ascending 60 degree: post-test | 10.63 (5.75)
  internal rotation ascending 90 degree: post-test | 11.29 (8.03)
  internal rotation ascending 120 degree: post-test | 13.25 (14.52)
  internal rotation descending 120 degree: pre-test | 12.52 (15.17)
  internal rotation descending 90 degree: pre-test | 12.66 (8.76)
  internal rotation descending 60 degree: pre-test | 11.95 (6.05)
  internal rotation descending 30 degree: pre-test | 11.28 (5.36)
  internal rotation descending 120 degree: post-test | 15.87 (14.88)
  internal rotation descending 90 degree: post-test | 13.66 (9.07)
  internal rotation descending 60 degree: post-test | 11.69 (6.50)
  internal rotation descending 30 degree: post-test | 10.86 (5.56)
  upward rotation ascending 30 degree: pre-test | 6.42 (3.66)
  upward rotation ascending 60 degree: pre-test | 18.88 (4.11)
  upward rotation ascending 90 degree: pre-test | 35.54 (4.84)
  upward rotation ascending 120 degree: pre-test | 52.78 (6.63)
  upward rotation ascending 30 degree: post-test | 6.29 (4.04)
  upward rotation ascending 60 degree: post-test | 19.34 (4.40)
  upward rotation ascending 90 degree: post-test | 36.51 (5.21)
  upward rotation ascending 120 degree: post-test | 54.35 (6.33)
  upward rotation descending 120 degree: pre-test | 53.92 (6.21)
  upward rotation descending 90 degree: pre-test | 38.10 (4.84)
  upward rotation descending 60 degree: pre-test | 21.18 (4.34)
  upward rotation descending 30 degree: pre-test | 7.34 (4.12)
  upward rotation descending 120 degree: post-test | 54.84 (6.29)
  upward rotation descending 90 degree: post-test | 38.44 (5.20)
  upward rotation descending 60 degree: post-test | 21.40 (4.73)
  upward rotation descending 30 degree: post-test | 7.01 (4.21)
Statistical Analysis 1: Comparison: Fatigued Group; The effects of muscle fatigue on scapular posterior tilt during scaption. Muscle fatigue would change scapular kinematics during scaption. Two way (angle x time) repeated measures. If there was an interaction between time and angle, further one way repeated measures would use to access the effects of time on kinematics changed of scapular posterior tilt during each angle of scaption; Test type: Other; p = 0.000467, ANOVA — The level of statistical significance was set at P < 0.05
Statistical Analysis 2: Comparison: Fatigued Group; The effects of time on kinematics changed of scapular posterior tilt during ascending 30 degree of scaption. One-way repeated measures analysis of variance; Test type: Other; p = 0.093, ANOVA — The level of statistical significance was adjusted at P<0.00625. (0.05/8=0.00625)
Statistical Analysis 3: Comparison: Fatigued Group; The effects of time on kinematics changed of scapular posterior tilt during ascending 60 degree of scaption. One-way repeated measures analysis of variance; Test type: Other; p = 0.062, ANOVA — The level of statistical significance was adjusted at P<0.00625. (0.05/8=0.00625)
Statistical Analysis 4: Comparison: Fatigued Group; The effects of time on kinematics changed of scapular posterior tilt during ascending 90 degree of scaption. One-way repeated measures analysis of variance; Test type: Other; p = 0.04, ANOVA — The level of statistical significance was adjusted at P<0.00625. (0.05/8=0.00625)
Statistical Analysis 5: Comparison: Fatigued Group; The effects of time on kinematics changed of scapular posterior tilt during ascending 120 degree of scaption. One-way repeated measures analysis of variance; Test type: Other; p = 0.000147, ANOVA — The level of statistical significance was adjusted at P<0.00625. (0.05/8=0.00625)
Statistical Analysis 6: Comparison: Fatigued Group; The effects of time on kinematics changed of scapular posterior tilt during descending 120 degree of scaption. One-way repeated measures analysis of variance; Test type: Other; p = 0.000012, ANOVA — The level of statistical significance was adjusted at P<0.00625. (0.05/8=0.00625)
Statistical Analysis 7: Comparison: Fatigued Group; The effects of time on kinematics changed of scapular posterior tilt during descending 90 degree of scaption. One-way repeated measures analysis of variance; Test type: Other; p = 0.007, ANOVA — The level of statistical significance was adjusted at P<0.00625. (0.05/8=0.00625)
Statistical Analysis 8: Comparison: Fatigued Group; The effects of time on kinematics changed of scapular posterior tilt during descending 60 degree of scaption. One-way repeated measures analysis of variance; Test type: Other; p = 0.059, ANOVA — The level of statistical significance was adjusted at P<0.00625. (0.05/8=0.00625)
Statistical Analysis 9: Comparison: Fatigued Group; The effects of time on kinematics changed of scapular posterior tilt during descending 30 degree of scaption. One-way repeated measures analysis of variance; Test type: Other; p = 0.032, ANOVA — The level of statistical significance was adjusted at P<0.00625. (0.05/8=0.00625)
Statistical Analysis 10: Comparison: Fatigued Group; The effects of muscle fatigue on scapular internal rotation during scaption Muscle fatigue would change scapular kinematics during scaption. Two way (angle x time) repeated measures. If there was an interaction between time and angle, further one way repeated measures would use to access the effects of time on kinematics changed of scapular internal rotation during each angle of scaption; Test type: Other; p = 0.000015, ANOVA — The level of statistical significance was set at P < 0.05
Statistical Analysis 11: Comparison: Fatigued Group; The effects of time on kinematics changed of scapular internal rotation during ascending 30 degree of scaption. One-way repeated measures analysis of variance; Test type: Other; p = 0.296, ANOVA — The level of statistical significance was adjusted at P<0.00625. (0.05/8=0.00625)
Statistical Analysis 12: Comparison: Fatigued Group; The effects of time on kinematics changed of scapular internal rotation during ascending 60 degree of scaption. One-way repeated measures analysis of variance; Test type: Other; p = 0.457, ANOVA — The level of statistical significance was adjusted at P<0.00625. (0.05/8=0.00625)
Statistical Analysis 13: Comparison: Fatigued Group; The effects of time on kinematics changed of scapular internal rotation during ascending 90 degree of scaption. One-way repeated measures analysis of variance; Test type: Other; p = 0.311, ANOVA — The level of statistical significance was adjusted at P<0.00625. (0.05/8=0.00625)
Statistical Analysis 14: Comparison: Fatigued Group; The effects of time on kinematics changed of scapular internal rotation during ascending 120 degree of scaption. One-way repeated measures analysis of variance; Test type: Other; p = 0.004, ANOVA — The level of statistical significance was adjusted at P<0.00625. (0.05/8=0.00625)
Statistical Analysis 15: Comparison: Fatigued Group; The effects of time on kinematics changed of scapular internal rotation during descending 120 degree of scaption. One-way repeated measures analysis of variance; Test type: Other; p = 0.002, ANOVA — The level of statistical significance was adjusted at P<0.00625. (0.05/8=0.00625)
Statistical Analysis 16: Comparison: Fatigued Group; The effects of time on kinematics changed of scapular internal rotation during descending 90 degree of scaption. One-way repeated measures analysis of variance; Test type: Other; p = 0.137, ANOVA — The level of statistical significance was adjusted at P<0.00625. (0.05/8=0.00625)
Statistical Analysis 17: Comparison: Fatigued Group; The effects of time on kinematics changed of scapular internal rotation during descending 60 degree of scaption. One-way repeated measures analysis of variance; Test type: Other; p = 0.636, ANOVA — The level of statistical significance was adjusted at P<0.00625. (0.05/8=0.00625)
Statistical Analysis 18: Comparison: Fatigued Group; The effects of time on kinematics changed of scapular internal rotation during descending 30 degree of scaption. One-way repeated measures analysis of variance; Test type: Other; p = 0.406, ANOVA — The level of statistical significance was adjusted at P<0.00625. (0.05/8=0.00625)
Statistical Analysis 19: Comparison: Fatigued Group; The effects of muscle fatigue on scapular upward rotation during scaption. Muscle fatigue would change scapular kinematics during scaption. Two way (angle x time) repeated measures. If there was an interaction between time and angle, further one way repeated measures would use to access the effects of time on kinematics changed of scapular upward rotation during each angle of scaption; Test type: Other; p = 0.001, ANOVA — The level of statistical significance was set at P < 0.05
Statistical Analysis 20: Comparison: Fatigued Group; The effects of time on kinematics changed of scapular upward rotation during ascending 30 degree of scaption. One-way repeated measures analysis of variance; Test type: Other; p = 0.650, ANOVA — The level of statistical significance was adjusted at P<0.00625. (0.05/8=0.00625)
Statistical Analysis 21: Comparison: Fatigued Group; The effects of time on kinematics changed of scapular upward rotation during ascending 60 degree of scaption. One-way repeated measures analysis of variance; Test type: Other; p = 0.141, ANOVA — The level of statistical significance was adjusted at P<0.00625. (0.05/8=0.00625)
Statistical Analysis 22: Comparison: Fatigued Group; The effects of time on kinematics changed of scapular upward rotation during ascending 90 degree of scaption. One-way repeated measures analysis of variance; Test type: Other; p = 0.021, ANOVA — The level of statistical significance was adjusted at P<0.00625. (0.05/8=0.00625)
Statistical Analysis 23: Comparison: Fatigued Group; The effects of time on kinematics changed of scapular upward rotation during ascending 120 degree of scaption. One-way repeated measures analysis of variance; Test type: Other; p = 0.005, ANOVA — The level of statistical significance was adjusted at P<0.00625. (0.05/8=0.00625)
Statistical Analysis 24: Comparison: Fatigued Group; The effects of time on kinematics changed of scapular upward rotation during descending 120 degree of scaption. One-way repeated measures analysis of variance; Test type: Other; p = 0.083, ANOVA — The level of statistical significance was adjusted at P<0.00625. (0.05/8=0.00625)
Statistical Analysis 25: Comparison: Fatigued Group; The effects of time on kinematics changed of scapular upward rotation during descending 90 degree of scaption. One-way repeated measures analysis of variance; Test type: Other; p = 0.389, ANOVA — The level of statistical significance was adjusted at P<0.00625. (0.05/8=0.00625)
Statistical Analysis 26: Comparison: Fatigued Group; The effects of time on kinematics changed of scapular upward rotation during descending 60 degree of scaption. One-way repeated measures analysis of variance; Test type: Other; p = 0.542, ANOVA — The level of statistical significance was adjusted at P<0.00625. (0.05/8=0.00625)
Statistical Analysis 27: Comparison: Fatigued Group; The effects of time on kinematics changed of scapular upward rotation during descending 30 degree of scaption. One-way repeated measures analysis of variance; Test type: Other; p = 0.263, ANOVA — The level of statistical significance was adjusted at P<0.00625. (0.05/8=0.00625)

5. Secondary Outcome: Change From Baseline in Scapular Muscle Activity During Shoulder Elevation in the Scapular Plane
Description: Test the ability of muscle activity (upper trapezius, lower trapezius, and serratus anterior) during shoulder elevation in the scapular plane (scaption).
  Muscle activation during scaption would divide into muscle activation during maximum voluntary isometric contraction (MVIC), present in percent.
Time Frame: through fatigue intervention completion, an average of 20 minutes in female subjects and 40 minutes in male subjects
Measure: Mean (Standard Deviation); unit: percentage of MVIC
Arm/Group | Fatigued Group
Number analyzed (Participants) | 30
percentage of MVIC
  serratus anterior ascending 30~60: pre-test | 40.65 (26.74)
  serratus anterior ascending 60~90: pre-test | 48.62 (38.33)
  serratus anterior ascending 90~120: pre-test | 65.91 (34.51)
  serratus anterior ascending 30~60: post-test | 51.38 (27.85)
  serratus anterior ascending 60~90: post-test | 62.70 (38.43)
  serratus anterior ascending 90~120: post-test | 84.61 (30.36)
  serratus anterior descending 120~90: pre-test | 30.88 (18.29)
  serratus anterior descending 90~60: pre-test | 23.03 (18.35)
  serratus anterior descending 60~30: pre-test | 13.99 (11.00)
  serratus anterior descending 120~90: post-test | 41.05 (17.06)
  serratus anterior descending 90~60: post-test | 29.09 (18.26)
  serratus anterior descending 60~30: post-test | 16.91 (12.04)
Statistical Analysis 1: Comparison: Fatigued Group; The effects of muscle fatigue on muscle activation of upper trapezius during scaption. Muscle fatigue would change muscle activation during scaption. Two way (angle x time) repeated measures. If there was an interaction between time and angle, further one way repeated measures would use to access the effects of time on muscle activation changed of upper trapezius during each angle of scaption; Test type: Other; p = 0.331, ANOVA — The level of statistical significance was set at P < 0.05
Statistical Analysis 2: Comparison: Fatigued Group; The effects of muscle fatigue on muscle activation of lower trapezius during scaption. Muscle fatigue would change muscle activation during scaption. Two way (angle x time) repeated measures. If there was an interaction between time and angle, further one way repeated measures would use to access the effects of time on muscle activation changed of lower trapezius during each angle of scaption; Test type: Other; p = 0.627, ANOVA — The level of statistical significance was set at P < 0.05
Statistical Analysis 3: Comparison: Fatigued Group; The effects of muscle fatigue on muscle activation of serratus anterior during scaption. Muscle fatigue would change muscle activation during scaption. Two way (angle x time) repeated measures. If there was an interaction between time and angle, further one way repeated measures would use to access the effects of time on muscle activation changed of serratus anterior during each angle of scaption; Test type: Other; p = 0.042, ANOVA — The level of statistical significance was set at P < 0.05
Statistical Analysis 4: Comparison: Fatigued Group; The effects of time on muscle activation changed of serratus anterior during ascending 30~60 degree of scaption. One-way repeated measures analysis of variance; Test type: Other; p = 0.021, ANOVA — The level of statistical significance was adjusted at P<0.0083. (0.05/6=0.0083)
Statistical Analysis 5: Comparison: Fatigued Group; The effects of time on muscle activation changed of serratus anterior during ascending 60~90 degree of scaption. One-way repeated measures analysis of variance; Test type: Other; p = 0.018, ANOVA — The level of statistical significance was adjusted at P<0.0083. (0.05/6=0.0083)
Statistical Analysis 6: Comparison: Fatigued Group; The effects of time on muscle activation changed of serratus anterior during ascending 90~120 degree of scaption. One-way repeated measures analysis of variance; Test type: Other; p = 0.002, ANOVA — The level of statistical significance was adjusted at P<0.0083. (0.05/6=0.0083)
Statistical Analysis 7: Comparison: Fatigued Group; The effects of time on muscle activation changed of serratus anterior during descending 120~90 degree of scaption. One-way repeated measures analysis of variance; Test type: Other; p = 0.002, ANOVA — The level of statistical significance was adjusted at P<0.0083. (0.05/6=0.0083)
Statistical Analysis 8: Comparison: Fatigued Group; The effects of time on muscle activation changed of serratus anterior during descending 90~60 degree of scaption. One-way repeated measures analysis of variance; Test type: Other; p = 0.035, ANOVA — The level of statistical significance was adjusted at P<0.0083. (0.05/6=0.0083)
Statistical Analysis 9: Comparison: Fatigued Group; The effects of time on muscle activation changed of serratus anterior during descending 60~30 degree of scaption. One-way repeated measures analysis of variance; Test type: Other; p = 0.05, ANOVA — The level of statistical significance was adjusted at P<0.0083. (0.05/6=0.0083)

6. Secondary Outcome: Change From Baseline in Scapular Muscle Recruitment Timing During Arm Elevation in Scapular Plane
Description: Test the ability of muscle onset timing (upper trapezius, lower trapezius, and serratus anterior) during shoulder elevation in the scapular plane (scaption).
  Onset timing was determined by EMG signals bigger than resting signals plus 3 times standard deviations.
  Origin was set at onset of kinematics data of glenohumeral joint.
Time Frame: through fatigue intervention completion, an average of 20 minutes in female subjects and 40 minutes in male subjects
Measure: Mean (Standard Deviation); unit: millisecond
Arm/Group | Fatigued Group
Number analyzed (Participants) | 30
millisecond
  upper trapezius: pre-test | -0.035 (0.326)
  lower trapezius: pre-test | 0.420 (0.563)
  serratus anterior: pre-test | -0.081 (0.204)
  upper trapezius: post-test | 0.004 (0.278)
  lower trapezius: post-test | 0.406 (0.560)
  serratus anterior: post-test | -0.05 (0.197)
Statistical Analysis 1: Comparison: Fatigued Group; The effects of muscle fatigue on muscle onset timing of upper trapezius during scaption. Muscle fatigue would change muscle onset timing during scaption. One-way repeated measures analysis of variance; Test type: Other; p = 0.5, ANOVA — The level of statistical significance was set at P < 0.05
Statistical Analysis 2: Comparison: Fatigued Group; The effects of muscle fatigue on muscle onset timing of lower trapezius during scaption. Muscle fatigue would change muscle onset timing during scaption. One-way repeated measures analysis of variance; Test type: Other; p = 0.843, ANOVA — The level of statistical significance was set at P < 0.05
Statistical Analysis 3: Comparison: Fatigued Group; The effects of muscle fatigue on muscle onset timing of serratus anterior during scaption. Muscle fatigue would change muscle onset timing during scaption. One-way repeated measures analysis of variance; Test type: Other; p = 0.466, ANOVA — The level of statistical significance was set at P < 0.05

ADVERSE EVENTS:
Time Frame: 1 year
Description: Collecting their reaction after fatigue task, and no one replied adverse event
Arm/Group | Fatigued Group
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-27): https://cdn.clinicaltrials.gov/large-docs/02/NCT03066102/Prot_SAP_000.pdf